CLINICAL TRIAL: NCT05797441
Title: Empowering Veterans to Self-Manage PTSD Symptoms Following Completion of Trauma-Focused Therapy
Brief Title: Testing the Effectiveness of a Therapist-Assisted Self-Management Program for Veterans Who Finished PTSD Therapy
Acronym: EMPOWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 20-102
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorders; PTSD; Self-Management
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Conducting a planning RCT in preparation for a fully powered trial using a parallel two-group pragmatic RCT design in which providers (n = 36) will be randomized at a 2:1 ratio to deliver either EMPOWER (n = 60) or TAU (n = 30) to veterans who have completed prolonged exposure or cognitive processing therapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMPOWER (Experimental): The goals of EMPOWER are to increase patients' self-efficacy for managing their PTSD, enable the maintenance or building upon gains made in TFT through the continued application of TFT skills, and encourage engagement in meaningful life activities. The program includes a Veteran workbook and four planned therapist contacts over the twelve weeks following TFT completion. The intervention includes: self-monitoring of symptoms, continued practice of TFT skills, engagement in meaningful activities, goal setting, and therapist support.
  Interventions: Behavioral: EMPOWER
- Treatment As Usual (Active Comparator): The comparison condition will be TAU following completion of TFT. In the spirit of TAU, providers will not be restricted in the type or intensity of services offered. Depending on local clinic policy or norms, providers randomized to TFT may provide post-TFT treatment themselves or Veterans may be referred to other providers and/or back to the clinician who referred the Veteran to TFT. If providers would have typically discharged Veterans following TFT, that is also allowable.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: EMPOWER — The goals of EMPOWER are to increase patients' self-efficacy for managing their PTSD, enable the maintenance or building upon gains made in TFT through the continued application of TFT skills, and encourage engagement in meaningful life activities. The program includes a Veteran workbook and four planned therapist contacts over the twelve weeks following TFT completion. The intervention includes: self-monitoring of symptoms, continued practice of TFT skills, engagement in meaningful activities, goal setting, and therapist support.
  Arms: EMPOWER
Other: Treatment As Usual — The comparison condition will be TAU following completion of TFT. In the spirit of TAU, providers will not be restricted in the type or intensity of services offered. Depending on local clinic policy or norms, providers randomized to TFT may provide post-TFT treatment themselves or Veterans may be referred to other providers and/or back to the clinician who referred the Veteran to TFT. If providers would have typically discharged Veterans following TFT, that is also allowable.
  Arms: Treatment As Usual

SUMMARY:
Patients who complete prolonged exposure and cognitive processing therapy, the treatments for posttraumatic stress disorder (PTSD) with the most empirical support, continue to express a need for mental health treatment. A therapist-assisted self-management program for patients who have completed one of these two treatments and achieved symptom improvement has the potential to meet patients' stated treatment needs, maintain or build upon their PTSD symptom reductions, increase their confidence in managing their symptoms, and reduce the number of mental health appointments that they need to attend. Further, reducing the number if mental health sessions attended by completers of these time and resource intensive psychotherapies will increase the likelihood that their implementation in regular-practice clinics will be maintained.

DETAILED DESCRIPTION:
Background. Nearly 90% of Veterans who complete trauma-focused therapy (TFT) for PTSD have remaining treatment needs. In the six-months following TFT, successful completers remain some of the highest utilizers of VA mental health services despite clinically meaningful symptom improvement. Prior work demonstrated that Veterans who benefitted from TFT's primary post-TFT treatment needs were the practice and application of skills learned during therapy, with the goal of maintaining or building upon treatment gains. Veterans expressed low self-efficacy for meeting these goals without the support of their therapists and feared stagnation or relapse without ongoing contact. As such, a therapist-assisted self-management program for TFT completers (EMPOWER) designed as a step down from active psychotherapy was developed and feasibility tested. The feasibility open trial demonstrated that EMPOWER is feasible and highly acceptable to patients. Further, findings suggest that the intervention was successful in helping Veterans maintain or enhance PTSD-related gains while reducing their mental health service utilization. These promising findings warrant a randomized evaluation.

Significance. Interventions that meet Veterans' post-TFT treatment needs are urgently needed. Mental health providers are delivering ongoing treatment to this high priority cohort of Veterans without evidence to guide their treatment plan. Further, higher than expected levels of post-TFT mental health care utilization threatens the continued implementation of these highly effective treatments. For all Veterans to have access to the most effective treatments for PTSD, interventions that prepare and enable successful TFT completers to step down from active therapy must evaluated and implemented.

Innovation. The proposed study is the first large-scale study of post-TFT care and the first to rigorously evaluate a self-management program to step-down from active to maintenance mental health services following a course of active psychotherapy.

Specific Aims: 1) Estimate posterior probability distributions of EMPOWER's effects and establish likely ranges for those effects as compared to post-TFT TAU for Veterans' MH service utilization and self-reported PTSD symptoms. The subsequent Hybrid RCT will be designed after assessing the likelihood of detecting an effect for EMPOWER across a range of sample sizes using Go/No Go and Overall Power methods. 2) Explore the impact of EMPOWER compared to post-TFT TAU on Veterans'(a) self-efficacy for managing PTSD symptoms, (b) satisfaction with post-TFT care, (c) well-being & functioning (d) depression, and (e) secondary utilization outcomes. 3) Conduct semi-structured interviews with Veterans and providers to contextualize quantitative findings and identify potential barriers, facilitators, and strategies to facilitate future implementation of EMPOWER.

Methodology: The study is a pragmatic randomized control trial (RCT) in which 36 PE and CPT providers will be randomized to support Veterans as they participate in the EMPOWER self-management program or facilitate TAU. Participants will be patients of the study providers who recently completed a course of PE/CPT during which they experienced clinically meaningful reductions in PTSD symptoms (n=90). Primary outcomes will be mental health service utilization (overall and with PE/CPT providers) and self-reported PTSD symptoms measured four times over a 9-month period. Qualitative interviews with providers (n=18) and Veterans (n=24) focused on providers' impressions of treatment effectiveness, implementation challenges/potential strategies, and Veterans' perception of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they:

  1. complete a course of individually-delivered TFT with a study therapist at a participating site
  2. experience a clinically meaningful change in PTSD symptomology
  3. at the time of enrollment (in either the TAU or EMPOWER arm), are not planning to initiate another weekly psychotherapy for PTSD for another mental or psychosocial condition within 3 months
  4. are willing to receive to either arm
  5. provide informed consent

Exclusion Criteria:

* Patients will be excluded if they report suicidal ideation that requires clinical monitoring at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist-5 (PCL-5) | 12 weeks post treatment initiation
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms
Veterans' Affairs Mental Health Service Utilization | 9 month period from treatment initiation to 9 months later
  All encounters with a mental health stop code in the Veterans Health Administration; variable is a count of total encounters
PTSD Checklist-5 (PCL-5) | 24 weeks post treatment initiation
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms
PTSD Checklist-5 (PCL-5) | 40 weeks post treatment initiation
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms

OTHER OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks post treatment initiation
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Client Satisfaction Questionnaire - 8 (CSQ-8) | 12 weeks post treatment initiation
  Treatment satisfaction; range = 8-32; higher scores = greater satisfaction
Brief Inventory of Psychosocial Functioning (BIPF) | 12 weeks post treatment initiation
  PTSD-related psychosocial functioning; higher scores = more functional impairment. Items are scored on a Likert scale from 0 (never) to 6 (always). Participants are instructed to skip any item that does not reflect a domain that they have participated in over the past 30 days. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100.
WHO Quality of Life, Brief (WHOQOL-BREF) | 12 weeks post treatment initiation
  Self-reported quality of life; higher score = better quality of life. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health. Subscales (domains): Physical Health (7 items) Psychological Health (6 items) Social Relationships (3 items) Environment (8 items) Scoring: Items scored 1-5. Raw domain score is the sum of respective item scores. All domain scores are then normalized to a range of 0-100. Refer to user manual for scoring algorithm.
Well-Being Inventory (WBI) | 12 weeks post treatment initiation
  The WBI is a multidimensional instrument that was designed to assess status, functioning, and satisfaction with four key life domains of vocation, finances, health, and social relationships. In total, there are 21 sections of the WBI and 126 questions/statements: 34 items for vocation, 24 for finances, 20 for health, and 48 for social relationships. Throughout the inventory, respondents are instructed to provide responses to categorical items (e.g., yes, no), or to endorse a single response from among statements using a 5-point Likert type response format (e.g., 1 = Never to 5 = Most or all of the time; 1 = Very dissatisfied to 5 = Very satisfied). Measures within each domain may be extracted from the full inventory and are available to use as separate entities depending on the needs of the administrator and/or the purpose of the assessment.
DSM-5 Cross-cutting symptom measure | 12 weeks post treatment initiation
  This measure assesses comorbid mental health conditions. The CCSM consists of 23 questions in a self-report format that evaluates mental health domains that are significant across psychiatric diagnoses. It is quick and easy to administer, taking patients around 5 minutes to complete in the waiting room. There are 13 psychiatric domains in this measure: depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. A 5-point scale (0-4) is used to record responses and reflect how much or how often the person has been concerned by a specific symptom over the previous 2 weeks. Additional inquiry is recommended if an individual scores a mild or slight rating, depending on the psychiatric symptom being investigated. This measure has good test-retest reliability in research settings and is useful and feasible in clinical practice.
Patient Health Questionnaire-9 (PHQ-9) | 24 weeks post treatment initiation
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Brief Inventory of Psychosocial Functioning (BIPF) | 24 weeks post treatment initiation
  PTSD-related psychosocial functioning; higher scores = more functional impairment. Items are scored on a Likert scale from 0 (never) to 6 (always). Participants are instructed to skip any item that does not reflect a domain that they have participated in over the past 30 days. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100.
WHO Quality of Life, Brief (WHOQOL-BREF) | 24 weeks post treatment initiation
  Self-reported quality of life; higher score = better quality of life. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health. Subscales (domains): Physical Health (7 items) Psychological Health (6 items) Social Relationships (3 items) Environment (8 items) Scoring: Items scored 1-5. Raw domain score is the sum of respective item scores. All domain scores are then normalized to a range of 0-100. Refer to user manual for scoring algorithm.
Well-Being Inventory (WBI) | 24 weeks post treatment initiation
  The WBI is a multidimensional instrument that was designed to assess status, functioning, and satisfaction with four key life domains of vocation, finances, health, and social relationships. In total, there are 21 sections of the WBI and 126 questions/statements: 34 items for vocation, 24 for finances, 20 for health, and 48 for social relationships. Throughout the inventory, respondents are instructed to provide responses to categorical items (e.g., yes, no), or to endorse a single response from among statements using a 5-point Likert type response format (e.g., 1 = Never to 5 = Most or all of the time; 1 = Very dissatisfied to 5 = Very satisfied). Measures within each domain may be extracted from the full inventory and are available to use as separate entities depending on the needs of the administrator and/or the purpose of the assessment.
DSM-5 Cross-cutting symptom measure | 24 weeks post treatment initiation
  This measure assesses comorbid mental health conditions. The CCSM consists of 23 questions in a self-report format that evaluates mental health domains that are significant across psychiatric diagnoses. It is quick and easy to administer, taking patients around 5 minutes to complete in the waiting room. There are 13 psychiatric domains in this measure: depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. A 5-point scale (0-4) is used to record responses and reflect how much or how often the person has been concerned by a specific symptom over the previous 2 weeks. Additional inquiry is recommended if an individual scores a mild or slight rating, depending on the psychiatric symptom being investigated. This measure has good test-retest reliability in research settings and is useful and feasible in clinical practice.
Patient Health Questionnaire-9 (PHQ-9) | 40 weeks post treatment initiation
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Brief Inventory of Psychosocial Functioning (BIPF) | 40 weeks post treatment initiation
  PTSD-related psychosocial functioning; higher scores = more functional impairment. Items are scored on a Likert scale from 0 (never) to 6 (always). Participants are instructed to skip any item that does not reflect a domain that they have participated in over the past 30 days. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100.
WHO Quality of Life, Brief (WHOQOL-BREF) | 40 weeks post treatment initiation
  Self-reported quality of life; higher score = better quality of life. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall QOL and general health. Subscales (domains): Physical Health (7 items) Psychological Health (6 items) Social Relationships (3 items) Environment (8 items) Scoring: Items scored 1-5. Raw domain score is the sum of respective item scores. All domain scores are then normalized to a range of 0-100. Refer to user manual for scoring algorithm.
Well-Being Inventory (WBI) | 40 weeks post treatment initiation
  he WBI is a multidimensional instrument that was designed to assess status, functioning, and satisfaction with four key life domains of vocation, finances, health, and social relationships. In total, there are 21 sections of the WBI and 126 questions/statements: 34 items for vocation, 24 for finances, 20 for health, and 48 for social relationships. Throughout the inventory, respondents are instructed to provide responses to categorical items (e.g., yes, no), or to endorse a single response from among statements using a 5-point Likert type response format (e.g., 1 = Never to 5 = Most or all of the time; 1 = Very dissatisfied to 5 = Very satisfied). Measures within each domain may be extracted from the full inventory and are available to use as separate entities depending on the needs of the administrator and/or the purpose of the assessment.
DSM-5 Cross-cutting symptom measure | 40 weeks post treatment initiation
  This measure assesses comorbid mental health conditions. The CCSM consists of 23 questions in a self-report format that evaluates mental health domains that are significant across psychiatric diagnoses. It is quick and easy to administer, taking patients around 5 minutes to complete in the waiting room. There are 13 psychiatric domains in this measure: depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. A 5-point scale (0-4) is used to record responses and reflect how much or how often the person has been concerned by a specific symptom over the previous 2 weeks. Additional inquiry is recommended if an individual scores a mild or slight rating, depending on the psychiatric symptom being investigated. This measure has good test-retest reliability in research settings and is useful and feasible in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M. Kehle-Forbes, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (8):
- United States (8):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05797441/ICF_000.pdf